CLINICAL TRIAL: NCT02334527
Title: Phase II Trial of Palbociclib (PD-0332991) in Patients With Metastatic Urothelial Cancer (UC) After Failure of First-Line Chemotherapy
Brief Title: Phase II Trial of Palbociclib in Patients With Metastatic Urothelial Cancer After Failure of First-Line Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Data from first 12 subjects-primary endpoint not met. Data analysis underway.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1406; 14-2196 (Other: UNC IRB)
Record Dates: First submitted 2015-01-06; First posted 2015-01-08 (Estimated); Results first posted 2018-04-24 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Metastatic Urothelial Carcinoma (UC)
Keywords: metastatic urothelial carcinoma (UC); LCCC 1406; Lineberger; palbociclib
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Palbociclib Single Arm trial (Other): Palbociclib
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — 125 mg capsule will be taken once per day orally and continuously for 3 weeks followed by 1 week off.
  Other Names: PD-0332991

SUMMARY:
This multicenter phase II trial will evaluate palbociclib (PD-0332991) in patients with metastatic urothelial carcinoma (UC) with cyclin-dependent kinase inhibitor 2A (CDKN2A) (also referred to as p16) loss and positive Retinoblastoma (Rb) expression after failure of first-line chemotherapy.

DETAILED DESCRIPTION:
This multicenter phase II trial will evaluate palbociclib (PD-0332991) in patients with metastatic urothelial carcinoma (UC) with cyclin-dependent kinase inhibitor 2A (CDKN2A) (also referred to as p16) loss and positive Retinoblastoma (Rb) expression after failure of first-line chemotherapy. The study will enroll up to 40 patients to identify 36 evaluable patients, using a Simon's two-stage design, with a primary endpoint of progression free survival (PFS) at 4 months (PFS4). Secondary objectives include estimating median PFS, overall survival (OS), response rate (RR) and exploratory objectives include an evaluation of molecular predictors of response and resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance status of ≤ 2 (see section 11.1, Appendix A)
* Histologically confirmed UC of the bladder, urethra, ureter or renal pelvis with Rb+/CDKN2A- based on immunohistochemistry (IHC) of tissue blocks or unstained slides performed within a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory at University of North Carolina (UNC); if stage I of original cohort indicates futility, molecular requirement for eligibility will change to Rb+/CCND1 overexpression (also based on IHC); see statistical section, section 8.0)
* Metastatic disease that is not amenable to curative surgery or radiation
* Prior treatment with ≤ two prior cytotoxic regimens; prior therapy must have consisted of at least one of the following: cisplatin, carboplatin, paclitaxel, docetaxel or gemcitabine. If the only prior cytotoxic therapy was administered in the perioperative i.e. neoadjuvant or adjuvant settings, patient is eligible provided the interval from end of therapy to the diagnosis of metastatic disease is less than one year.
* Progressive disease during or after treatment with at least one of the agents listed above
* At least one measurable disease site (as defined by Response Evaluation Criteria In Solid Tumors (RECIST)1.1) that has not been previously irradiated
* No prior therapy with a CDK 4/6 inhibitor; prior anti PD-1 and anti PD-L1 therapy is permitted
* Washout period should be at least 2 weeks for prior chemotherapy or radiation therapy 3.1.10 Resolution of all acute toxic effects of prior chemotherapy, radiotherapy, surgery to ≤ grade 1 per NCI Common Terminology Criteria for Adverse Events (CTCAE)v4 except neuropathy which may be ≤ grade 2
* No active brain metastases
* Adequate bone marrow, liver and renal functions as assessed by the following:

  * Hemoglobin ≥ 8 g/dL;
  * Absolute neutrophil count ≥ 1,500/uL;
  * Platelets ≥ 75,000 g/uL;
  * Total bilirubin ≤ 1.5 times upper limit of normal (ULN);
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN;
  * serum creatinine ≤ 2.5 times ULN;
* Negative serum pregnancy test in women of child-bearing potential within 7 days of D1 of treatment
* If fertile, agree to use effective contraception (condom or other barrier methods, oral contraceptives, implantable contraceptives, intrauterine devices) during trial
* Life expectancy greater than 3 months
* Subject must be able to give written Institutional Review Board (IRB) approved informed consent and be able to follow protocol requirements

Exclusion Criteria:

* Any prior treatment with any investigational drug within the preceding 4 weeks
* Any concurrent active malignancy requiring treatment (other than basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, superficial bladder tumors, other malignancies curatively treated > 3 years prior to study entry) or patients with adenocarcinoma of the prostate that has been surgically treated and with a post-treatment prostate-specific antigen (PSA) that is non-detectable.
* Unstable systemic disease or active uncontrolled infection
* Major surgery, open biopsy or significant traumatic injury within 4 weeks prior to study entry
* Not willing to avoid grapefruit, grapefruit juices, grapefruit hybrids, Seville oranges, pomelos, and exotic citrus fruits from 7 days prior to the dose of study medication and during the entire study due to potential CYP3A4 interaction with the study medication. Orange juice is allowed.
* Intake of any herbal preparations or medications (including, but not limited to, Saint John's Wort and ginkgo biloba) and dietary supplements within 7 days prior to first dose of study drug
* Unable or unwilling to discontinue use of any drug known to be a strong or moderate inhibitor or inducer of CYP3A4 (prohibited inducers and inhibitors must be discontinued within 2 weeks prior to first dose of study drug; see section 11.2 Appendix B); unable or unwilling to discontinue use of any proton pump inhibitor; see section 11.2, Appendix B
* Any malabsorption problem that, in the investigator's opinion, would prevent adequate absorption of the study drug
* Inability to swallow oral medications
* Pregnant or breast-feeding
* Substance abuse, or medical, psychological or social conditions that may interfere with the patient's participation in the study or the evaluation of the study results
* Other serious, ongoing, non-malignant disease or infection that would compromise protocol objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-03-17 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2017-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew I Milowsky, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (3):
- United States (3):
  - University of Michigan, Ann Arbor, Michigan
  - North Carolina Cancer Hospital (UNC), Chapel Hill, North Carolina
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center — http://cancer.med.unc.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 12 patients were enrolled between April 2015 and January 2017.
Pre-assignment Details: 34 patients were screened, 25 were eligible based on tumor immunohistochemistry (IHC) demonstrating p16 loss and intact retinoblastoma. Of those, 12 patients were enrolled.
Groups:
- Palbociclib (Single Arm Trial): Palbociclib
  Palbociclib: 125 mg capsule will be taken once per day orally and continuously for 3 weeks followed by 1 week off.
Period: Overall Study
Arm/Group | Palbociclib (Single Arm Trial)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm (Single Arm Trial): Palbociclib
  Palbociclib: 125 mg capsule will be taken once per day orally and continuously for 3 weeks followed by 1 week off.
Arm/Group | Single Arm (Single Arm Trial)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 68 [51 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 10
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Primary Tumor Site [Count of Participants; unit: Participants]
  Bladder | 7
  Upper Tract | 4
  Urethra | 1
Number of prior systemic therapy regiments (including immunotherapy) [Count of Participants; unit: Participants]
  1 | 7
  2 | 3
  3 | 2
Setting of prior platinum-based chemotherapy [Count of Participants; unit: Participants]
  Perioperative only | 8
  Metastatic only | 2
  Both | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — Measure Description: A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  Participants
    0 | 5
    1 | 6
    2 | 1
Hemoglobin [Count of Participants; unit: Participants]
  <10 g/dL | 2
  >= 10 g/dL | 10
Liver Metastases [Count of Participants; unit: Participants]
  Yes | 0
  No | 12
Time from prior therapy [Count of Participants; unit: Participants]
  < 3 months | 4
  3-6 months | 5
  6-9 months | 1
  >=12 months | 2

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Estimate progression free survival (PFS) at 4 months in patients with metastatic urothelial cancer (UC) who have progressed after first-line chemotherapy. PFS is defined as the percent of patients who are alive and free from progression at 4 months.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm (Single Arm Trial)
Number analyzed (Participants) | 12
Participants | 2

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from D1 of treatment until progression or death as a result of any cause. Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: 4 Months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib Single Arm Trial
Number analyzed (Participants) | 12
Months | 1.9 [1.8 to 3.7]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from day 1 of treatment until death as a result of any cause.
Time Frame: Patients will be followed for up to 5 years after removal from study therapy or death, whichever occurs first.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Palbociclib (Single Arm Trial)
Number analyzed (Participants) | 12
Months | 6.3 [2.2 to 12.6]

4. Secondary Outcome: Response Rate (RR) - Total Number of Patients With Complete Response (CR) and/or Partial Response (PR)
Description: Estimate response rate (RR) in patients with metastatic UC who have progressed after first-line chemotherapy. Response rate will be the number of patients with complete response and/or partial response. Response will be based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Radiographic response will be measured by RECIST, Response Evaluation Criteria In Solid Tumors Criteria, indicating if subject experienced a Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), no response or less response than Partial or Progressive; or Progressive Disease (PD), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 4 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Palbociclib (Single Arm Trial)
Number analyzed (Participants) | 12
Participants | 0

5. Secondary Outcome: Number of Participants With Adverse Events
Description: Characterize the safety profile of palbociclib in patients with metastatic UC after first-line chemotherapy. The NCI Common Terminology Criteria for Adverse Events is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Groups:
- Any Grade Adverse Events; Grade >=3 Adverse Event: Palbociclib
  Palbociclib: 125 mg capsule will be taken once per day orally and continuously for 3 weeks followed by 1 week off.
Arm/Group | Any Grade Adverse Events | Grade >=3 Adverse Event
Number analyzed (Participants) | 12 | 12
Participants
  Any Adverse Event | 12 | 11
  Any Treatment Related Adverse Event | 11 | 9

ADVERSE EVENTS:
Time Frame: 32 weeks
Arm/Group | Single Arm (Single Arm Trial)
All-Cause Mortality (participants affected / at risk) | 11/12
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (Single Arm Trial) (N=12)
Confusion (Psychiatric disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (Single Arm Trial) (N=12)
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase increased (Investigations) | 2
Anemia (Blood and lymphatic system disorders) | 10
Anorexia (Metabolism and nutrition disorders) | 1
Aspartate aminotransferase increased (Investigations) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Constipation (Gastrointestinal disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
General disorders and administration site conditions - Other, specify (General disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 5
Lymphocyte count decreased (Investigations) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 8
Pain (General disorders) | 2
Platelet count decreased (Investigations) | 5
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Renal hemorrhage (Renal and urinary disorders) | 1
Right Mid-Back Pain (General disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Weight loss (Investigations) | 2
White blood cell decreased (Investigations) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days